CLINICAL TRIAL: NCT04408274
Title: Remediation of Emotional Deficits in Multiple Sclerosis and Traumatic Brain Injury: A Piolt Study
Brief Title: Remediation of Emotional Deficits in Multiple Sclerosis and Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jean Lengenfelder, Associate Director, Traumatic Brain Injury Lab, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-764-13
Record Dates: First submitted 2018-04-17; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis; Traumatic Brain Injury
Keywords: Processing Speed; Intervention; Multiple Sclerosis; Traumatic Brain Injury; Cognition
MeSH Terms: conditions — Multiple Sclerosis; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized Tests (Experimental)
  Interventions: Behavioral: Emotional Processing Training
- Placebo Control (Placebo Comparator)
  Interventions: Behavioral: Placebo Control

INTERVENTIONS:
Behavioral: Emotional Processing Training
  Arms: Computerized Tests
Behavioral: Placebo Control
  Arms: Placebo Control

SUMMARY:
This study will examine the efficacy of a clinical intervention for improving emotional processing in individuals with MS and TBI.(1)The main outcome measure will be changes in emotional processing measures from pre to post treatment.

(2)This study will also assess the impact of the emotional processing intervention on changes in pre and post treatment depression and anxiety, as well as fatigue.(3) This study will additionally measure the impact of the emotional processing intervention on cognitive functioning, specifically processing speed, attention and executive abilities. This will be accomplished through the completion of a neuropsychological battery prior to and following the completion of treatment.(4)Finally, the investigators will measure the impact of the intervention on quality of life and social functioning, utilizing a pre and post treatment assessment consisting of measures of self-efficacy, quality of life, functional abilities, and awareness.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Multiple Sclerosis or Traumatic Brain Injury
* Fluent in English
* processing speed impairment (based on evaluation)

Exclusion Criteria:

* currently taking steroids and/or benzodiazepines
* prior stroke or neurological diease
* history of significant pyschiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Epilepsy, Bipolar Disorder
* significant alcohol or drug abuse history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in scores on Facial Expression Identification Task (FEIT) | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  The FEIT assesses one's ability to correctly identify and discriminate emotions from faces

SECONDARY OUTCOMES:
Change in scores on Emotion Regulation Questionnaire (ERQ) | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  The ERQ is a self-report measure of the use of 2 emotional regulation strategies: cognitive reappraisal and expressive suppression
Change in scores on Satisfaction with Life Scale (SWLS) | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  The SWLS is a self-report measure of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States